CLINICAL TRIAL: NCT04201132
Title: Protection Against Emboli During Carotid Artery Stenting Using a 3-in-1 Delivery System Comprised of a Post-dilation Balloon, Integrated Embolic Filter and a Novel Carotid Stent - the PERFORMANCE II Study
Brief Title: Protection Against Emboli During Carotid Artery Stenting Using the Neuroguard IEP System
Acronym: PERFORMANCE II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Contego Medical, Inc. (Industry)
Collaborators: Yale Cardiovascular Research Group (Other); Advance Research Associates (Other); CardioMed Device Consultants, LLC (Industry); Iqvia Pty Ltd (Industry); Medidata Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP1400
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Carotid Artery Stenosis; Carotid Artery Diseases; Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Carotid artery stenting (Experimental): Carotid artery stenting procedure with Neuroguard IEP System
  Interventions: Device: Carotid artery stenting with Neuroguard IEP System

INTERVENTIONS:
Device: Carotid artery stenting with Neuroguard IEP System — Carotid artery stenting (treatment) with the Neuroguard IEP 3-in-1 Carotid Stent and Post-Dilation Balloon System with Integrated Embolic Protection

SUMMARY:
A prospective, multicenter single-arm, open label study to evaluate the safety and effectiveness of the Neuroguard IEP System for the treatment of carotid artery stenosis in subjects at elevated risk for adverse events following carotid endarterectomy (CEA).

DETAILED DESCRIPTION:
The Neuroguard IEP System is a 3-in-1 carotid stent delivery system consisting of an angioplasty balloon, an integrated embolic protection device and a nitinol self-expanding stent loaded over the balloon and constrained by an outer sheath. Eligible patients must be between 20 and 80 years of age and diagnosed with either de-novo atherosclerotic or post CEA restenotic lesion(s) in the internal carotid arteries (ICA) or at the carotid bifurcation with ≥50% stenosis if symptomatic), or, ≥80% stenosis if asymptomatic (both defined by angiography using NASCET methodology). Symptomatic patients are defined as having stroke or TIA ipsilateral to the carotid lesion within 180 days of the procedure within the hemisphere supplied by the target vessel. Enrolled subjects will be followed at 30 days, 6 months, 12 months, 24 months and 36 months.

ELIGIBILITY:
General Inclusion Criteria

1. Male and non-pregnant, non-breastfeeding female subjects whose age is ≥ 20 years and ≤ 80.
2. Patient is willing and capable of complying with all study protocol requirements, including the specified follow-up visits and can be contacted by telephone.
3. Patient or his/her authorized legal representative must sign a written informed consent form that has been approved by the local governing Institutional Review Board (IRB)/ Ethics Committee (EC) of the respective clinical site.
4. Patient is diagnosed with carotid artery stenosis treatable with carotid artery stenting and is considered a high operative risk for CEA.
5. Patient is diagnosed with either:

   1. Symptomatic carotid stenosis ≥ 50% as determined by angiography using NASCET methodology. Symptomatic is defined as ipsilateral transient monocular blindness: amaurosis fugax; ipsilateral carotid transient ischemic attack (TIA), with neurologic symptoms persisting less than 24 hours; or ipsilateral non-disabling stroke within 180 days of the procedure; or
   2. Asymptomatic carotid stenosis ≥ 80% as determined by angiography using NASCET methodology.
6. Patient has a modified Rankin Scale score of ≤ 2 at the time of informed consent.
7. Females of child-bearing potential have a negative pregnancy test within 24 hours of the index procedure.
8. Patient is willing and able to take dual antiplatelet therapy for a minimum of 30 days following the index procedure.

Angiographic Inclusion Criteria

1. Target lesion located at the carotid bifurcation and/or proximal internal carotid artery (ICA).
2. Single de novo or restenotic (post carotid endarterectomy (CEA)) target lesion or severe tandem lesions that can be covered by a single Neuroguard stent.
3. Target lesion length is ≤ 20 mm (for 30 mm stents) or is ≤ 30 mm (for 40 mm stents).
4. Index vessel diameter (segment covered by the mid-portion of the stent) between 4.0 mm and 6.0 mm at the site of the target lesion.
5. Distal vessel diameter at the site of filter deployment is between 4.0 mm to 7.0 mm.
6. Distal common carotid artery diameter (segment covered by proximal portion of the stent) is between 4.0 mm and 8.0 mm
7. Sufficient landing zone exists in the cervical internal carotid artery distal to the target lesion to allow for the safe and successful deployment of both the primary embolic protection filter and the Neuroguard filter.

High Risk for CEA Conditions For inclusion in the study, a patient must meet at least one significant anatomic or comorbid high risk conditions listed below. Patients at high risk for CEA are defined as having significant comorbidities and/or anatomic risk factors and would be poor candidates for carotid endarterectomy (CEA) in the opinion of a physician.

High Anatomic Risk for CEA Conditions

1. Target lesion at or above C2 (level of jaw) or below the clavicle.
2. Inability to extend the head due to cervical arthritis or other cervical disorders.
3. History of radiation treatment to the neck or radical neck dissection
4. Prior head and neck surgery in the region of the carotid artery.
5. Spinal immobility of the neck.
6. Tracheostomy or tracheostoma.
7. Hostile neck or surgically inaccessible lesion
8. Laryngeal palsy or laryngectomy.
9. Severe tandem lesions (total length must be ≤ 30 mm and must be covered with one stent).
10. Occlusion of the contralateral CCA or ICA.
11. Severe bilateral ICA stenosis.

High Co-morbid Risk Conditions for CEA

1. Patient is ≥ 70 years of age (maximum 80 years) at the time of enrollment.
2. NYHA Class III or IV congestive heart failure (CHF)
3. Chronic obstructive pulmonary disease (COPD) with FEV1 < 50 or on intermittent or chronic oxygen therapy.
4. Left ventricular ejection fraction (LVEF) ≤ 35%
5. Unstable angina
6. History of recent MI (between 14 days and 6 weeks prior to index the procedure)
7. Coronary artery disease with two or more vessels with ≥ 70% stenosis
8. Planned coronary artery bypass grafting (CABG) or valve replacement surgery between 31 and 60 days after CAS procedure
9. Peripheral vascular surgery or abdominal aortic aneurysm repair is required and planned between 31 and 60 days following CAS procedure
10. Contralateral laryngeal nerve paralysis
11. Restenosis following a prior carotid endarterectomy (CEA).

General Exclusion Criteria:

1. Life expectancy of less than one year, cancer with metastatic spread, undergoing active chemotherapy treatment, or currently requiring an organ transplantation.
2. An evolving acute stroke.
3. Anticipated or potential sources of emboli including left ventricular aneurysm, severe cardiomyopathy, aortic or mitral mechanical heart valve, severe calcific aortic stenosis (valve area < 1.0 cm2), endocarditis, moderate to severe mitral stenosis, known previously symptomatic PFO, left atrial thrombus, any intracardiac mass or DVT or PE treated within the past 12 months.
4. History of paroxysmal atrial flutter or atrial fibrillation requiring chronic anticoagulation
5. History of chronic atrial flutter or atrial fibrillation.
6. Anticoagulation with Phenprocoumon (Marcumar®), warfarin, or a direct thrombin inhibitor, or anti-Xa agents within 14 days of the index procedure.
7. Acute febrile illness (temperature > 100.4F or 38C) or active infection.
8. Subjects with presumptive or confirmed SARS-CoV-2/COVID-19 infection.

   * A SARS-CoV-2/COVID-19 test shall be performed 72 hours prior to the index procedure for all subjects
   * Note: If a subject has confirmed SARS-CoV-2/COVID-19 infection (SARSCoV-2/COVID-19+), eligibility may be re-established 21 days following diagnosis if infection is asymptomatic and 21 days following resolution of symptoms if infection is symptomatic.
9. Acute myocardial infarction < 14 days prior to index procedure.
10. Any major surgical procedure (i.e. intraabdominal or intrathoracic surgery or any surgery / interventional procedure involving cardiac or vascular system) 30 days prior to or following the index procedure.
11. History of major disabling stroke with substantial residual disability (modified Rankin score ≥ 3)
12. Known severe carotid stenosis or complete occlusion contralateral to the target lesion requiring treatment within 30 days of the index procedure.
13. Other neurological deficit not due to stroke that may confound the neurological assessments.
14. Dementia considered other than mild.
15. Known hypersensitivity to nitinol or its components (e.g. nickel, titanium).
16. History of intracranial hemorrhage within 90 days prior to the index procedure.
17. History of GI bleed within 30 days prior to the index procedure
18. Chronic renal insufficiency (serum creatinine ≥ 2.5 ml/dL or estimated GFR < 30 cc/min)
19. Any condition that precludes proper angiographic assessment or makes percutaneous arterial access unsafe (e.g., severe hepatic impairment, malignant hypertension, morbid obesity).
20. Known hypersensitivity to contrast media that cannot be adequately premedicated.
21. Hemoglobin (Hgb) < 8 gm/dL, platelet count < 100,000, INR > 1.5 (irreversible), or heparin-induced thrombocytopenia.
22. History or current indication of bleeding diathesis or coagulopathy including thrombocytopenia or an inability to receive heparin in amounts sufficient to maintain an activated clot time at ≥ 250 seconds.
23. Contraindication to standard of care study medications, including antiplatelet therapy or aspirin.
24. Currently enrolled in another interventional device or drug study that has not yet reached the primary endpoint.
25. Potential for subject non-compliance with protocol-required follow up or anti platelet medication in the opinion of the investigator.

Angiographic Exclusion Criteria

1. Total occlusion of the target carotid artery.
2. Previously placed stent in the ipsilateral carotid artery.
3. Severe calcification or vascular tortuosity of the target vessel that may preclude the safe introduction of the sheath, guiding catheter, distal filter, Neuroguard stent or Neuroguard filter. Excessive circumferential calcification of the target lesion is defined as >3 mm of thickness of calcification seen in orthogonal views on fluoroscopy. Severe vascular tortuosity is defined as 2 or more bends of 90 degrees or more within 4 cm of the target lesion.
4. Qualitative characteristics of stenosis and stenosis-length of carotid bifurcation (common carotid) and/or ipsilateral external carotid artery, that preclude the safe introduction of the sheath.
5. Angulation or tortuosity (≥ 90 degree) of the innominate and common carotid artery (CCA) that precludes safe, expeditious sheath placement or that will transmit a severe loop to the internal carotid after sheath placement.
6. Angiographic evidence of a mobile filling defect or fresh thrombus in the target carotid artery.
7. Presence of "string sign" of the target lesion (a sub-totally occluded, long segment of the true lumen of the artery with markedly reduced contrast flow).
8. Non-atherosclerotic carotid stenosis (e.g. dissection, fibromuscular dysplasia)
9. Proximal/ostial CCA, innominate stenosis, or intracranial stenosis located distal to the target stenosis that is more severe that target stenosis.
10. Patient in whom percutaneous vascular access is not possible, including severe tortuosity or stenosis that requires additional endovascular procedures to facilitate aortic arch access or that prevents safe and expeditious access.
11. Patient with intracranial pathology that, in the opinion of the investigator, makes the patient inappropriate for study participation (e.g., arteriovenous malformations, brain tumor, microangiopathy or large vessel cerebral vascular disease, etc) or that would confound the neurological evaluation.
12. Known mobile plaque or thrombus in the aortic arch.
13. Type III aortic arch.
14. Angiographic, CT, MR or ultrasound evidence of severe atherosclerosis, tortuosity or angulation of the aortic arch or origin of the innominate or common carotid arteries that would preclude or make difficult safe passage of the sheath and other endovascular devices to the target artery as needed for carotid stenting.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MAE | 30 days
  Death, all stroke and myocardial infarction (MI)
Ipsilateral Stroke | 12 months
  Ipsilateral hemiparesis

SECONDARY OUTCOMES:
Technical success | Day of procedure
  Successful stent deployment, successful filter deployment and retrieval, successful stent post-dilation and successful delivery system retrieval
Procedure success | Day of procedure
  Successful stent implantation with <50% residual stenosis
TLR | 12 months
  Target Lesion Revascularization
In-Stent Restenosis (ISR) | 12 months, 24 months, 36 months
  Restenosis of stented segment
Major stroke | 30 days
  New focal ischemic neurological deficit of abrupt onset which is present after 7 days and results in greater than or equal to 4 point increase in NIHSS compared to baseline.
Minor stroke | 30 days
  New focal ischemic neurological deficit of abrupt onset lasting > 24 hours and increases NIHSS by less than or equal to 3 points at 7 days
Transient Ischemic Attack (TIA) | 30 days
  Focal ischemic neurological deficit of abrupt onset and of presumed vascular etiology that resolves completely within 24 hours of onset
Neurological death | 12 months
  Death after a stroke that is either a direct consequence of the stroke or a complication of the stroke

CONTACTS AND LOCATIONS:
Overall Officials: William A Gray, MD, Principal Investigator — Main Line Health; Ralf Langhoff, MD, Principal Investigator — Sankt Gertrauden Krankenhaus
Locations (38):
- United States (28):
  - Huntsville Hospital, Huntsville, Alabama
  - St. Helena Hospital, St. Helena, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Manatee Memorial Hospital, Bradenton, Florida
  - Lyerly Baptist Neurosurgery, Jacksonville, Florida
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Lexington, Lexington, Kentucky
  - Terrebonne General Medical Center, Houma, Louisiana
  - White Oak Medical Center, Silver Spring, Maryland
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University at Buffalo Neurosurgery, Buffalo, New York
  - Mt. Sinai, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - North Carolina Heart and Vascular Research, Raleigh, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - St. Vincent Hospital, Erie, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Harrisburg, Pennsylvania
  - Lankenau Institute, Wynnewood, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Prisma Health Midlands, Columbia, South Carolina
  - Prisma Health Upstate, Greenville, South Carolina
  - Monument Health - Rapid City Regional Hospital, Rapid City, South Dakota
  - North Central Heart Institute, Sioux Falls, South Dakota
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - Ballad Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Turkey Creek Medical Center, Knoxville, Tennessee
  - Texas Heart Institute, Houston, Texas
- Acibadem City Clinic University Hospital, Sofia, Bulgaria
- Germany (6):
  - University Herzzentrum Bad Krozingen, Bad Krozingen
  - Sankt Gertrauden-Krankenhaus GmbH, Berlin
  - Cardiovascular Centre Frankfurt, Frankfurt
  - Medizinisches Versorgungszentrum Prof. Mathey, Prof. Schofer GmbH, Hamburg
  - Universitätsklinikum Leipzig, Leipzig
  - Elblandklinikum Radebeul, Radebeul
- Centro Cardiologico Monzino, Milan, Italy
- University Clinic of Cardiology Skopje, Skopje, North Macedonia
- University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gray WA, Metzger DC, Zidar J, Kedev S, Petrov I, Soukas P, Levy E, Bachinsky W, Bacharach JM, Montorsi P, Novack V, Lansky A, Langhoff R. The PERFORMANCE II Trial: A Prospective Multicenter Investigation of a Novel Carotid Stent System. JACC Cardiovasc Interv. 2025 Feb 10;18(3):367-376. doi: 10.1016/j.jcin.2024.10.031. Epub 2025 Jan 8. PMID 39797836